CLINICAL TRIAL: NCT05257421
Title: The Immediate Effect Of Shockwave Therapy On the Quadratus Lumborum (QL) Muscle Trigger Points vs Regular Back Exercises in Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: The Immediate Effect Of Shockwave Therapy On the Quadratus Lumborum (QL) Muscle Trigger Points vs Regular Back Exercises in Chronic Nonspecific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Maram Mohammed Taha Makki, physiotherapist / master student, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWTQLRCT2022
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- shockwave group (Experimental)
  Interventions: Device: shockwave machine
- exercise group (Active Comparator)
  Interventions: Other: leg and back exercises
- combined group (Active Comparator)
  Interventions: Combination Product: shockwave and exercises

INTERVENTIONS:
Device: shockwave machine — shockwave therapy. 2000 impulses will be applied, 1000 on the TrPs and 1000 surrounding it, with Energy level up to 2,5 bars and frequency of 10Hz
  Arms: shockwave group
Other: leg and back exercises — the exercise program will include 5 exercises that focuses on the back and lower limbs. These exercises are:
  * Bridge
  * Plank
  * Squat
  * Push-ups
  * Back extension Each exercise will be done for 3-5 sets.
  Arms: exercise group
Combination Product: shockwave and exercises — both types of interventions will be applied for the patient
  Arms: combined group

SUMMARY:
the study aims to compare the effect of regular back exercises with shockwave therapy by treating male patients with non-specific low back pain between the age of (20-40). Who will be devided into 3 groups, and will be treated by shockwave therapy , exercises or both combined. After signing a consent form, patients will be assigned to the groups blindly, so the patients will not know if they are in the experimental or control group.

Hypothesis:

The hypothesis of this study states that:

o Research hypothesis: there will be a significant difference between the radial ESWT and back exercises in reducing LBP

ELIGIBILITY:
Inclusion Criteria:

* Only male patients will be included.
* Age 20-40 years old.
* Non-specific LBP for at least 3 months.
* At least one local tenderness or active trigger point in the anatomical region of the QL muscle.
* Pain intensity on numerical pain scale should be more than 4

Exclusion Criteria:

* LBP due to a pathology or trauma.
* Below 20 years of age.
* Previous lumbar surgeries.
* Malignancy.
* Patients under medications or painkillers.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
pressure-pain threshold | 45 hour session
  Algometry device will be used to measure three thresholds' values:
  * Tenderness threshold.
  * Referred pain threshold.
  * Pain tolerance threshold.
The Oswestry Disability Index | 45 minutes session
  is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability, scoring from 0 to 50, the lower score the better
Numerical pain scale | 45 minutes session
  0-10 the lower the better

SECONDARY OUTCOMES:
ROM of the back | 45 minutes session
  an electrical goniometer will be used to measure the change in the back ROM

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Epidemiological features of chronic low-back pain
- [Background] Joshi S, Sheth M. Effect of extracorporeal shockwave therapy on myofascial pain syndrome of upper trapezius: A systematic review. Int J Med Sci Public Health. 2020;9(10):1.
- [Background] Effect of Static Versus Dynamic Ultrasound on Pain in Subjects with Trigger Point in Quadratus Lumborum Having Non-Specific Chronic Low Back. 2020;10(December):263-9.